CLINICAL TRIAL: NCT00517933
Title: Sildenafil Trial of Exercise Performance in Idiopathic Pulmonary Fibrosis
Acronym: STEP-IPF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00018538; U10HL080413 (NIH); 507
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Fibrosis; Hypertension, Pulmonary
Keywords: Idiopathic Pulmonary Fibrosis; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary; Idiopathic Pulmonary Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): 20 mg of sildenafil 3 times a day (TID) for 12 weeks followed by 20 mg of sildenafil TID for an additional 12 weeks
  Interventions: Drug: Sildenafil Citrate
- Placebo / Sildanafil (Placebo Comparator): 20 mg of placebo TID for 12 weeks followed by 20 mg of sildenafil citrate TID for an additional 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — Sildenafil citrate (20mg 3 times a day [TID] orally for 12 weeks followed by 20mg TID open-label sildenafil for an additional 12 weeks)
  Other Names: Revatio
  Arms: Sildenafil
Other: Placebo — Placebo (20mg TID orally for 12 weeks followed by 20mg open-label sildenafil for 12 weeks)
  Arms: Placebo / Sildanafil

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease that affects an individual's ability to breathe. This study will evaluate the effectiveness of sildenafil, a medication that increases blood flow to the lungs, at improving breathing function, exercise capacity, and quality of life in people with advanced IPF.

DETAILED DESCRIPTION:
IPF is a disease in which fibrous tissue clogs the lungs. This eventually damages air sacs in the lungs and leads to widespread and permanent scarring of lung tissue. Individuals with IPF may experience breathing difficulties, cough, chest pain, and a decreased exercise capacity. Pulmonary hypertension, which is high blood pressure in the arteries of the lungs, affects half of all people with IPF. The fibrous tissue that clogs the lungs also blocks blood from flowing through the lungs effectively, reducing the amount of oxygen in the lungs. The fibrous tissue also reduces the lungs' ability to use what oxygen is available. These factors can cause breathing difficulties and may eventually lead to heart disease. Sildenafil is a medication that can increase blood supply to the lungs and reduce the heart's workload. The purpose of this study is to evaluate the effectiveness of sildenafil at improving breathing function, exercise capacity, and quality of life in people with advanced IPF.

This study will enroll people with advanced IPF. Participants will be randomly assigned to receive sildenafil or placebo three times a day for 12 weeks. Study visits will occur at baseline and Weeks 1, 6, and 12. At Week 12, participants will have the option to continue in the study for an additional 12 weeks. All participants who agree to continue in the study will receive sildenafil three times a day for the second 12 weeks. Study visits will occur at Weeks 13, 18, and 24. At all study visits, a physical exam and blood collection will occur. At selected visits, the following study procedures will occur: lung function testing; urine collection; a 6-minute walk test, which will measure the distance walked in a 6-minute period; and questionnaires to assess health status, breathing, and quality of life. Participants will record medication usage and symptoms in a daily diary. Study researchers will review medical records and the Social Security death index 5 years following the end of the study to determine the incidence of death among study participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IPF
* Diffusing capacity of the lung (DLCO) level less than 35% (adjusted for hemoglobin)

Exclusion Criteria:

* Current enrollment in another investigational study
* Six-minute walk distance of less than 50 meters at screening or study entry
* Difference of greater than 15% between the screening and study entry 6-minute walk distance
* Acute or long-term impairment other than dyspnea (e.g., angina pectoris, intermittent claudication) that limits the ability to comply with the 6-minute walk test or other study requirements
* Forced Expiratory Volume 1-second (FEV1)/forced vital capacity (FVC) ratio of less than 0.65 after bronchodilator use
* Extent of emphysema greater than the extent of fibrotic change (e.g., honeycombing, reticular changes) on high-resolution computed tomography (HRCT) scan
* Acute heart attack within the 6 months prior to study entry
* Nitrate use
* Hypersensitivity to sildenafil or any component of the formulation
* Presence of aortic stenosis (AS)
* Life-threatening arrhythmia within 1 month of study entry
* Diabetes mellitus requiring insulin therapy
* Second-degree or third-degree atrioventricular (AV) block on electrocardiogram
* Severe chronic heart failure, defined by left ventricular ejection fraction (LVEF) of less than 25%
* Presence of idiopathic hypertrophic subaortic stenosis (IHSS)
* Hypotension (i.e., systolic blood pressure [SBP] less than 100 mm Hg or diastolic blood pressure [DBP] less than 50 mm Hg)
* Uncontrolled systemic hypertension (i.e., SBP greater than 180 mm Hg or DBP greater than 100 mm Hg)
* Known penile deformities or conditions (e.g., sickle cell anemia, multiple myeloma, leukemia) that may predispose participant to priapism
* Aspartate aminotransferase (AST), serum glutamic pyruvic transaminase (SGPT), alanine aminotransferase (ALT), or serum glutamic oxaloacetic transaminase (SGOT) greater than three times the upper limit of normal range
* Kidney impairment (i.e., creatinine clearance less than 30 mL/minute)
* Current drug or alcohol dependence
* Retinitis pigmentosa
* History of vision loss
* History of nonarteritic ischemic optic neuropathy
* Recently initiated pulmonary rehabilitation within 30 days of study entry. Participants will be prohibited from starting pulmonary rehabilitation during the study. Participants who are currently undergoing maintenance pulmonary rehabilitation at study entry will be asked to maintain their levels of rehabilitation for the duration of the study.
* Use of any investigational therapy as part of a clinical trial for any medical condition within 30 days of study entry
* Start or change in dose of treatment for IPF investigational agent (e.g., interferon gamma-1b, pirfenidone, etanercept, N-acetylcysteine, any other investigational agent intended to treat IPF), corticosteroids, or cytotoxic agents within 30 days of study entry
* Use of certain medications. More information about this criterion can be found in the study protocol.
* Treatment for pulmonary hypertension with prostaglandins (e.g., epoprostenol, treprostinil), endothelin-1 antagonists (e.g., bosentan, sitaxsentan, ambrisentan), or any other phosphodiesterase inhibitor (e.g., tadalafil, vardenafil) within 30 days of study entry
* Addition or discontinuation of calcium channel blockers, digitalis, diuretics, or vasodilators within 30 days of study entry (dosage must be stable for 7 days prior to study entry [except for diuretics])
* Currently on the waiting list for a lung transplant
* Use of L-arginine supplements
* Use of grapefruit juice or St. John's wort
* Pregnant or breastfeeding
* Resting saturation of peripheral oxygen (SpO2) (i.e., oxygen saturation measured using pulse oximetry) less than 92% with 6 liters of supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hunninghake, MD, Study Chair — University of Iowa; Kevin Brown, MD, Principal Investigator — National Jewish Health; Rob Kaner, MD, Principal Investigator — Weill Medical College at Cornell University; Talmadge King, MD, Principal Investigator — University of California, San Francisco; Joe Lasky, MD, Principal Investigator — Tulane University; James Loyd, MD, Principal Investigator — Vanderbilt University; Fernando Martinez, MD, Principal Investigator — University of Michigan; Imre Noth, MD, Principal Investigator — University of Chicago; Ganesh Raghu, MD, Principal Investigator — University of Washington; Jesse Roman, MD, Principal Investigator — Emory University; Jay Ryu, MD, Principal Investigator — Mayo Clinic; David Zisman, MD, Principal Investigator — University of California, Los Angeles; Kevin Anstrom, PhD, Principal Investigator — Duke University; Herbert Reynolds, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Lake D Morrison, MD, Principal Investigator — Duke University
Locations (13):
- United States (13):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Andrade J, Schwarz M, Collard HR, Gentry-Bumpass T, Colby T, Lynch D, Kaner RJ; IPFnet Investigators. The Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet): diagnostic and adjudication processes. Chest. 2015 Oct;148(4):1034-1042. doi: 10.1378/chest.14-2889. PMID 26111071
- [Derived] Durheim MT, Collard HR, Roberts RS, Brown KK, Flaherty KR, King TE Jr, Palmer SM, Raghu G, Snyder LD, Anstrom KJ, Martinez FJ; IPFnet investigators. Association of hospital admission and forced vital capacity endpoints with survival in patients with idiopathic pulmonary fibrosis: analysis of a pooled cohort from three clinical trials. Lancet Respir Med. 2015 May;3(5):388-96. doi: 10.1016/S2213-2600(15)00093-4. Epub 2015 Apr 15. PMID 25890798
- [Derived] Idiopathic Pulmonary Fibrosis Clinical Research Network; Zisman DA, Schwarz M, Anstrom KJ, Collard HR, Flaherty KR, Hunninghake GW. A controlled trial of sildenafil in advanced idiopathic pulmonary fibrosis. N Engl J Med. 2010 Aug 12;363(7):620-8. doi: 10.1056/NEJMoa1002110. Epub 2010 May 18. PMID 20484178
- See also: Click here for the Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet) Web site — http://www.ipfnet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil / Sildenafil: 20 mg oral sildenafil 3 times per day
- Placebo / Sildenafil: 20 mg oral placebo 3 times per day
Period: Period 1
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Started | 89 (Patients decreased due to death, adverse event, lost to follow up and other (see below)) | 91 (Patients decreased due to death, adverse event and other (see below))
Completed | 81 | 85
Not Completed | 8 | 6
Not completed — Death | 2 | 1
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Underwent lung transplant | 0 | 1
Period: Period 2
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Started | 79 (2 patients terminated after completion of period one, but before starting period 2) | 83 (2 patients terminated after completion of period one, but before starting period 2)
Completed | 73 | 70
Not Completed | 6 | 13
Not completed — Death | 2 | 4
Not completed — Adverse Event | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Underwent lung transplant | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: 20 mg of oral sildenafil 3 times per day for 12 weeks, followed by 20 mg oral sildenafil 3 times per day for 12 weeks
- Placebo: 20 mg of placebo 3 times per day for 12 weeks, followed by 20 mg open-label sildenafil 3 times per day for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.7) | 68.2 (9.3) | 69.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 75 | 75 | 150
Region of Enrollment [Number; unit: participants]
  United States | 89 | 91 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Distance From Enrollment to Week 12 (≥ 20% Improvement)
Description: This is a binary score (1 or 0) with 1 being better than 0. All models adjust for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Measured at Week 12
Measure: Number; unit: participants
Groups:
- Sildenafil: 20 mg of oral sildenafil 3 times per day for 12 weeks, followed by 20 mg oral sildenafil 3 times per day for an additional 12 weeks.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
participants | 9 | 6
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.39, Chi-squared

2. Secondary Outcome: 6-minute Walk Distance (6MWT)
Description: The 6MWT measures the distance that a participant can walk in a period of 6 minutes.
Time Frame: Baseline, 6 week, 12 week
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
meters
  1st baseline | 246.93 (99.11) | 267.71 (127.75)
  2nd baseline | 246.39 (103.40) | 269.55 (129.83)
  6 week | 237.29 (121.48) | 257.55 (139.44)
  12 week | 239.09 (126.39) | 249.48 (138.46)

3. Secondary Outcome: Estimated Change From Baseline to 12 Weeks in 6-minute Walk Distance
Description: The 6MWT measures the distance that a participant can walk in a period of 6 minutes. All models adjust for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, week 12
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
meters | -28.5 [-43.2 to -13.8] | -45.2 [-59.7 to -30.8]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.11, Regression, Linear; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [-3.9 to 37.3]

4. Secondary Outcome: Desaturation During 6-minute Walk Test (6MWT)
Description: The 6MWT was stopped when the pulse oximetry (SpO2) dropped to below 80% for six consecutive seconds. The estimates are based on the Kaplan-Meier event curves with minutes walked as the x-axis.
Time Frame: Week 12
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Number analyzed (Participants) | 89 | 91
percentage of participants | 83.6 [74.4 to 91.0] | 75.3 [65.3 to 84.3]
Statistical Analysis 1: Comparison: Sildenafil / Sildenafil vs Placebo / Sildenafil; Test type: Superiority or Other; p = 0.41, Log Rank

5. Secondary Outcome: Change in Dyspnea
Description: The University of California at San Diego Shortness of Breath Questionnaire (SOBQ) uses a 6-point scale (0 = "not at all" to 5 = "maximal or unable to do because of breathlessness") to rate 24 items. The final score ranges from 0 to 120 -- lower scores are better.
Time Frame: Measured from enrollment to 12 weeks (phase I)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | 0.22 [-3.10 to 3.54] | 6.81 [3.53 to 10.08]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Slope = -6.58, 95% CI 2-sided [-11.25 to -1.92], Standard Error of Mean 2.3

6. Secondary Outcome: University of California at San Diego (UCSD) Shortness of Breath Questionnaire Total
Description: The University of California at San Diego Shortness of Breath Questionnaire (SOBQ) uses a 6-point scale (0 = "not at all" to 5 = "maximal or unable to do because of breathlessness") to rate 24 items. The final score ranges from 0 to 120 -- lower scores are better. (Raw scores)
  Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 50.71 (22.00) | 43.28 (20.18)
  6 week | 49.67 (22.74) | 47.64 (25.61)
  12 Week | 50.58 (23.41) | 48.13 (24.10)
  Change from Baseline to 6 weeks | -1.27 (12.63) | 4.42 (17.16)
  Change from Baseline to 12 weeks | 0.30 (16.01) | 6.99 (18.43)

7. Secondary Outcome: Change in Forced Vital Capacity (FVC) Adjusted Values
Description: Change in FVC (liters) from baseline (time 0) to week 12 comparing the sildenafil and placebo groups. Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, Week 12
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Number analyzed (Participants) | 89 | 91
liters | -0.04 [-0.09 to -0.00] | -0.05 [-0.10 to -0.01]
Statistical Analysis 1: Comparison: Sildenafil / Sildenafil vs Placebo / Sildenafil; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.05 to 0.07]

8. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Raw scores of FVC (liters) from baseline (time 0) to week 6 and 12 comparing the sildenafil and placebo groups
Time Frame: Baseline, Week 6, Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Number analyzed (Participants) | 89 | 91
liters
  Baseline | 2.25 (0.70) | 2.42 (0.75)
  Week 6 | 2.25 (0.72) | 2.40 (0.74)
  Week 12 | 2.22 (0.75) | 2.36 (0.78)
  Change from baseline to 6 weeks | -0.03 (0.21) | -0.03 (0.15)
  Change from baseline to 12 weeks | -0.04 (0.23) | -0.05 (0.20)

9. Secondary Outcome: Change in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) Adjusted Values
Description: Change in DLCO (% predicted) measured at baseline (time 0), and week 12 comparing the sildenafil and placebo groups. All models adjust for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, Week 12
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted (DLCO)
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Number analyzed (Participants) | 89 | 91
percentage of predicted (DLCO) | -0.30 [-1.4 to 0.7] | -1.9 [-2.9 to -0.8]
Statistical Analysis 1: Comparison: Sildenafil / Sildenafil vs Placebo / Sildenafil; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [0.1 to 3.0]

10. Secondary Outcome: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: Raw scores of DLCO (% predicted) measured at baseline (time 0), week 6, and week 12 comparing the sildenafil and placebo groups
Time Frame: Baseline, Week 6, Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of predicted (DLCO)
Arm/Group | Sildenafil / Sildenafil | Placebo / Sildenafil
Number analyzed (Participants) | 89 | 91
percentage of predicted (DLCO)
  Baseline | 25.81 (6.03) | 26.73 (6.16)
  Week 6 | 26.00 (7.05) | 26.11 (6.28)
  Week 12 | 25.66 (6.79) | 25.38 (7.43)
  Change from baseline to 6 weeks | -0.07 (4.35) | -1.15 (4.59)
  Change from baseline to 12 weeks | -0.33 (4.58) | -1.78 (6.32)

11. Secondary Outcome: Change in Borg Dyspnea Index (BDI) After 6 Minute Walk Test (Adjusted Values)
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum) and indicates the degree of breathlessness after completion of the 6-minute walk test. Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 week
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | 0.04 [-0.30 to 0.37] | 0.37 [0.04 to 0.70]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.16, Regression, Linear; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.81 to 0.14]

12. Secondary Outcome: Borg Dyspnea Index (BDI) After 6 Minute Walk Test (Raw Scores)
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum) and indicates the degree of breathlessness after completion of the 6-minute walk test.
Time Frame: Baseline, 6 week, 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 3.72 (1.79) | 3.23 (1.80)
  6 week | 3.53 (1.91) | 3.42 (1.79)
  12 week | 3.76 (2.22) | 3.49 (1.61)
  Change from Baseline to 6 week | -0.23 (1.37) | 0.37 (1.42)
  Change from Baseline to 12 week | 0.09 (1.62) | 0.39 (1.70)

13. Secondary Outcome: Change in St. George's Respiratory Questionnaire (Total Score) (Adjusted Values)
Description: The St. George's Respiratory Questionnaire asks patients how breathing problems impair their life and is scored from 0 (no impairment) to 100 (maximum impairment.) Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 week
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -1.6 [-3.9 to 0.6] | 2.5 [0.2 to 4.7]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.01, Regression, Linear; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-7.3 to -0.9]

14. Secondary Outcome: St. George's Respiratory Questionnaire (Total Score)
Description: Mean raw scores of the St. George's Respiratory Questionnaire. The St. George's Respiratory Questionnaire asks patients how breathing problems impair their life and is scored from 0 (no impairment) to 100 (maximum impairment.)
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 54.55 (16.46) | 51.72 (15.86)
  6 week | 52.56 (16.81) | 51.74 (16.45)
  12 Week | 52.58 (16.35) | 52.19 (16.26)
  Change from Baseline to 6 weeks | -1.45 (10.11) | 1.65 (10.53)
  Change from Baseline to 12 weeks | -1.71 (12.35) | 2.88 (10.61)

15. Secondary Outcome: Change in St. George's Respiratory Questionnaire (Symptoms Score) Adjusted Value
Description: The St. George's Respiratory Questionnaire asks patients how breathing problems impair their life and is scored from 0 (no impairment) to 100 (maximum impairment). Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -3.6 [-7.0 to -0.1] | 2.2 [-1.3 to 5.6]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.02, Regression, Linear; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-10.6 to -0.9]

16. Secondary Outcome: St. George's Respiratory Questionnaire (Symptoms Score)
Description: The St. George's Respiratory Questionnaire asks patients how breathing problems impair their life and is scored from 0 (no impairment) to 100 (maximum impairment). Mean raw scores of the St. George's Respiratory Questionnaire. Mean raw scores of the St. George's Respiratory Questionnaire.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 58.20 (17.75) | 53.99 (18.90)
  6 week | 55.89 (17.72) | 56.26 (18.77)
  12 Week | 54.49 (17.59) | 55.55 (19.08)
  Change from Baseline to 6 weeks | -2.05 (16.72) | 3.15 (16.30)
  Change from Baseline to 12 weeks | -3.57 (17.95) | 2.80 (14.74)

17. Secondary Outcome: Change in St. George's Respiratory Questionnaire (Activity Score) Adjusted Value
Description: as for outcome 15
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -1.2 [-3.7 to 1.4] | 2.5 [0.0 to 5.0]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.04, Regression, Linear; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-7.2 to -0.1]

18. Secondary Outcome: St. George's Respiratory Questionnaire (Activity Score)
Description: The St. George's Respiratory Questionnaire asks patients how breathing problems impair their life and is scored from 0 (no impairment) to 100 (maximum impairment). Mean raw scores of the St. George's Respiratory Questionnaire.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 71.20 (17.50) | 68.02 (17.63)
  6 week | 69.95 (18.66) | 67.44 (18.51)
  12 Week | 69.75 (18.63) | 69.13 (19.34)
  Change from Baseline to 6 weeks | -1.95 (10.82) | 0.28 (10.87)
  Change from Baseline to 12 weeks | -1.25 (12.56) | 2.77 (13.27)

19. Secondary Outcome: Change in St. George's Respiratory Questionnaire (Impacts Score) Adjusted Value
Description: as for outcome 15
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -0.9 [-3.8 to 2.0] | 2.8 [-0.0 to 5.7]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-7.8 to 0.4]

20. Secondary Outcome: St. George's Respiratory Questionnaire (Impacts Score)
Description: as for outcome 18
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 43.20 (19.26) | 39.77 (18.81)
  6 week | 41.62 (19.49) | 41.58 (19.68)
  12 Week | 41.95 (19.23) | 41.05 (18.81)
  Change from Baseline to 6 weeks | -0.67 (12.79) | 2.37 (12.94)
  Change from Baseline to 12 weeks | -0.91 (15.90) | 3.15 (13.11)

21. Secondary Outcome: Change in ICECAP-O Adjusted Value
Description: The ICEpop CAPability measure for Older people (ICECAP-O) is a measure of capability in older people for use in economic evaluation. The values of ICECAP-O range from 0 (worst) to 1 (best).
  Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | 0.00 [-0.02 to 0.03] | -0.02 [-0.04 to 0.00]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.18, Regression, Linear; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.06]

22. Secondary Outcome: ICECAP-O
Description: The ICEpop CAPability measure for Older people (ICECAP-O) is a measure of capability in older people for use in economic evaluation. The values of ICECAP-O range from 0 (worst) to 1 (best). Mean raw scores of ICECAP-O.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 0.79 (0.14) | 0.81 (0.13)
  6 week | 0.80 (0.16) | 0.76 (0.17)
  12 Week | 0.79 (0.14) | 0.81 (0.14)
  Change from Baseline to 6 weeks | 0.02 (0.12) | -0.05 (0.12)
  Change from Baseline to 12 weeks | 0.00 (0.11) | -0.02 (0.10)

23. Secondary Outcome: Change in EuroQOL Thermometer (Adjusted Value)
Description: The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate a better health state.
  Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | 0.5 [-3.1 to 4.1] | -1.8 [-5.3 to 1.7]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.37, Regression, Linear; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-2.8 to 7.3]

24. Secondary Outcome: EuroQOL Thermometer
Description: The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate a better health state.
  Mean raw scores of EuroQOL Thermometer.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 66.49 (17.45) | 67.66 (16.98)
  6 week | 69.47 (16.92) | 67.09 (19.65)
  12 Week | 66.96 (16.45) | 67.05 (16.37)
  Change from Baseline to 6 weeks | 2.51 (15.32) | -1.40 (17.23)
  Change from Baseline to 12 weeks | 0.49 (17.28) | -2.12 (19.08)

25. Secondary Outcome: Change in EuroQOL (EQ-5D) Utility - Adjusted Value
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in total score range -0.594 to 1.000; higher score indicates better health state.
  Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -0.01 [-0.06 to 0.03] | -0.03 [-0.08 to 0.01]

26. Secondary Outcome: EuroQOL (EQ-5D) Utility
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in total score range -0.594 to 1.000; higher score indicates better health state.
  Mean raw scores of EuroQOL Utility.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 0.71 (0.24) | 0.74 (0.19)
  6 week | 0.75 (0.23) | 0.71 (0.25)
  12 Week | 0.70 (0.26) | 0.72 (0.21)
  Change from Baseline to 6 weeks | 0.04 (0.18) | -0.02 (0.24)
  Change from Baseline to 12 weeks | -0.01 (0.23) | -0.03 (0.19)

27. Secondary Outcome: Change in Short Form Health Survey (SF36) General Health - Adjusted Value
Description: The SF36 measures functional health and well-being scores on eight scales that correlate with two aggregate scores.
  Each score ranges from 0 to 100, with a higher score indicating better function.
  Values adjusted for baseline values of age, height, sex, white race, and DLCO. Values from models are estimated changes from baseline to 12 weeks (with 95% confidence intervals). The difference estimate is based on sildenafil - placebo.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -1.0 [-2.5 to 0.4] | -3.9 [-5.4 to -2.4]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.008, Regression, Linear; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [0.8 to 5.0]

28. Secondary Outcome: Short Form Health Survey (SF36) General Health
Description: The SF36 measures functional health and well-being scores on eight scales that correlate with two aggregate scores.
  Each score ranges from 0 to 100, with a higher score indicating better function.
  Mean raw scores of SF36 General Health
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | 36.99 (9.64) | 37.66 (8.73)
  6 week | 36.00 (9.85) | 34.97 (8.64)
  12 Week | 36.31 (8.91) | 34.39 (8.41)

29. Secondary Outcome: Change in SF36 Aggregate Physical (Adjusted Value)
Description: as for outcome 27
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale | -0.5 [-1.9 to 0.8] | -0.4 [-1.7 to 1.0]
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.86, Regression, Linear; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.7]

30. Secondary Outcome: Short Form Health Survey (SF36) Aggregate Physical
Description: The SF36 measures functional health and well-being scores on eight scales that correlate with two aggregate scores.
  Each score ranges from 0 to 100, with a higher score indicating better function.
  Mean raw scores of SF36 Aggregate Physical.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 89 | 91
units on a scale
  Baseline | -1.68 (0.92) | -1.52 (0.87)
  6 week | -1.70 (0.99) | -1.58 (0.91)
  12 Week | -1.71 (0.86) | -1.51 (0.89)
  Change from Baseline to week 6 | -0.06 (0.52) | -0.08 (0.64)
  Change from Baseline to week 12 | -0.05 (0.56) | -0.05 (0.63)

ADVERSE EVENTS:
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 13/89 | 15/91
Other Adverse Events (participants affected / at risk) | 72/89 | 62/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=89) | Placebo (N=91)
Respiratory, thoracic, or mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (11)
Infection or infestation (Infections and infestations) | 3 (4) | 2 (2)
Cardiac disorder (Cardiac disorders) | 1 (1) | 3 (3)
GI disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Colitis ischemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=89) | Placebo (N=91)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 13 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 7 (8)
Bronchitis (Infections and infestations) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 18 (22) | 17 (19)
Dizziness (Nervous system disorders) | 8 (9) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 8 (8)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Oedema peripheral (General disorders) | 9 (11) | 8 (9)
Hypotension (Vascular disorders) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Findings are limited to patients with advanced IPF. It is unknown if treatment effect was driven by particular subgroup of patients. Study was too short and enrolled too few to assess duration of effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No